CLINICAL TRIAL: NCT00152932
Title: Ocular Blood Flow Measured by HRF and CLBF in Newly Diagnosed and Early Glaucoma Patients Before and After Instillation of Dorzolamide 2%
Brief Title: Ocular Blood Flow in Early Glaucoma Patients Before and After Treatment With Dorzolamide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 04-0645-A
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2005-09

CONDITIONS: Glaucoma
Keywords: Glaucoma; Intraocular pressure; Ocular blood flow; Laser-Doppler Flowmetry
MeSH Terms: conditions — Glaucoma | interventions — dorzolamide

INTERVENTIONS:
Drug: Dorzolamide 2% drops
Device: HRF and CLBF

SUMMARY:
Impaired ocular blood flow is an important risk factor in the pathogenesis of primary open angle glaucoma (POAG). A few studies suggest that topical dorzolamide 2% may increase optic nerve perfusion. The objectives of this study are to learn the effects of dorzolamide on the retinal and optic nerve blood flow of glaucoma patients.

The present study is a prospective, randomized, double-masked, crossover design study of newly diagnosed or already treated patients with early glaucoma.

The investigators will check ocular blood flow parameters using the Canon Laser Blood Flowmeter (CLBF), used to evaluate retinal arteriole blood flow, and the Heidelberg retinal flowmeter (HRF), which measures blood flow through capillary beds in the retina and optic nerve head.

Any demonstrated improvements to retinal and optic nerve blood flow with dorzolamide, will mean that the drug may protect against ischaemic nerve and retinal damage. Any documented improvement in flow could lead to a major change in the management of glaucoma patients as well as other retinal ischemic diseases such as diabetic retinopathy and central retinal vein occlusion.

DETAILED DESCRIPTION:
High intraocular pressure (IOP) is the major risk factor for glaucoma. Lowering intraocular pressure is still the only accepted form of treatment for glaucoma.

Over the past decade, epidemiological and experimental evidence suggested that impaired ocular blood flow is an important risk factor with an important role in the pathogenesis of primary open angle glaucoma (POAG). Several studies suggest that ischemia-promoting vascular factors may contribute to glaucomatous damage including vasospasm, impaired ocular perfusion pressure and general vascular disorders such as low blood pressure, especially dips in blood pressure at night.

Different techniques are employed to assess vascular dysfunction in the eye. As the methodology of ocular blood flow assessment is complex and differs in various aspects (e.g. target tissue and physiological parameters), comparative studies are required in order to enhance the interpretation of these measurements.

Our laboratory has state of the art equipment to assess ocular blood flow. One study done by us suggested that one drop of Dorzolamide 2% does not improve retinal blood flow in normal eyes. In the present study we plan to extend this study to 2 weeks of treatment in patients with POAG.

Dorzolamide hydrochloride 2% is a topical carbonic anhydrase inhibitor which reduces intraocular pressure (IOP) by decreasing the production of aqueous humour. Pharmacological studies on volunteers and glaucoma patients, using Color Doppler Imaging (measuring the retrobulbar blood flow) and Scanning laser Ophthalmoscopy (measuring arteriovenous passage time), indicate that topically applied Dorzolamide may increase perfusion of the optic nerve and peripapillary retina.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 20-80 years of age.
2. Presence of typical early glaucomatous optic disc changes (cup/disc ratio ≤ 0.75) and/or early glaucomatous visual field defects (mean deviation less than 5dB and outside of 10° from fixation) in the study eye at the baseline visit.
3. Best corrected visual acuity of at least 20/40.
4. Signed informed consent from the subject
5. The subject should be able to understand the instructions and perform the HRF and CLBF tests as well as be willing and able to comply with the study schedule and treatment.

Exclusion Criteria:

1. Pregnant women or nursing mothers.
2. Any other active ocular disease (ocular infections, Uveitis, etc.)
3. Known allergy or sensitivity to the study medications.
4. Functionally significant visual field loss (mean deviation greater than 5dB) or cup/disc ratio greater than 0.75 or evidence of progressive visual field loss within the last 6 months.
5. Required chronic use of other ocular or systemic hypotensive medications during the study, other than the study medication (e.g. beta-blockers, Ca-channel blockers)
6. Vascular occlusive disease affecting the ocular circulation such as: diabetic retinopathy, central retinal vein occlusion, central retinal artery occlusion, or non-arteritic ischemic optic neuropathy.
7. Previous intraocular surgery or ocular traumas.
8. Any past history of serious systemic condition affecting cerebral circulation including: hypertension, diabetes, cerebral vascular accident (CVA), or coronary artery bypass graft (CABG).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2005-05; Study Completion 2006-06

PRIMARY OUTCOMES:
Ocular blood flow measurements

SECONDARY OUTCOMES:
Intraocular pressure reduction

CONTACTS AND LOCATIONS:
Overall Officials: Graham E Trope, MB, FRCSC, Principal Investigator — University of Toronto, Department of Ophthalmology; Chris Hudson, PhD, Study Chair — Department of Ophthalmology, Toronto Western Hospital, Toronto; John Flanagan, PhD, Study Chair — Department of Ophthalmology, Toronto Western Hospital, Toronto; Yvonne M Buys, MD, FRCSC, Study Chair — University of Toronto, Department of Ophthalmology, Toronto Western Hospital, Toronto
Locations (1):
- Department of Ophthalmology and Visual Sciences; Toronto Western Hospital, Toronto, Ontario, Canada